CLINICAL TRIAL: NCT07313618
Title: Safety and Efficacy of a Single Suprachoroidal Injection of JWK010 Gene Therapy in Subjects With Oculocutaneous Albinism Type 1 (OCA1)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Fang Lu, Professor, West China Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-1619
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Oculocutaneous Albinism (OCA)
Keywords: TYR gene; OCA1
MeSH Terms: conditions — Albinism, Oculocutaneous

STUDY DESIGN:
Intervention Model Description: This study employs a traditional '3+3' dose escalation design. It is planned to enroll up to 3 dose cohorts. Each cohort will initially enroll 3 participants. Based on the observed dose-limiting toxicities, a cohort may be expanded to include 6 participants. Therefore, the anticipated total sample size for this study ranges from 9 to 18 participants. The enrollment number provided in this registration (18) represents the maximum possible number of participants to be enrolled.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- JWK010 at Dose 1 (Experimental): Suprachoroidal injection dose 1 of JWK010 in one eye
  Interventions: Genetic: JWK010 gene therapy
- JWK010 at Dose 2 (Experimental): Suprachoroidal injection dose 2 of JWK010 in one eye
  Interventions: Genetic: JWK010 gene therapy
- JWK010 at Dose 3 (Experimental): Suprachoroidal injection dose 3 of JWK010 in one eye
  Interventions: Genetic: JWK010 gene therapy

INTERVENTIONS:
Genetic: JWK010 gene therapy — JWK010: AAV vector containing a coding sequence for tyrosinase.

SUMMARY:
Oculocutaneous albinism (OCA) is the most common type of albinism. People with OCA have little or no pigment (melanin) in their eyes, skin, and hair. This often leads to symptoms such as sensitivity to light, crossed or misaligned eyes, reduced vision, and involuntary eye movements.

OCA type 1 is caused by changes in the tyrosinase gene, which results in a lack or reduced function of the tyrosinase enzyme. This enzyme is essential for producing melanin, so people with OCA1 cannot make enough of it.

JWK010 is a gene therapy product developed specifically for patients with OCA1. It is designed to help the cells produce functional tyrosinase protein, with the goal of restoring pigment in the retina and improving retinal structure and function.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the purpose and requirements of this trial, voluntarily participate in the clinical study and sign the informed consent form (for minor subjects, the informed consent form shall be signed by their guardians), and be able to cooperate with all required tests according to the study protocol.
2. Aged ≥5 years and ≤12years (inclusive of the threshold values, based on the date of signing the informed consent form), regardless of gender.
3. Clinically diagnosed with OCA1A type, with ocular and cutaneous manifestations consistent with the clinical presentation of OCA1A.
4. Confirmed by genetic testing to carry pathogenic mutations in both TYR alleles, without carrying pathogenic mutations associated with other ophthalmic genetic diseases.
5. The visual acuity of the fellow eye is better than that of the study eye, and the visual acuity of the fellow eye is no less than 20/400

Exclusion Criteria:

1. Presence of any other condition in the study eye that may cause vision loss (e.g., optic atrophy, advanced glaucoma, uveitis).
2. The presence of lens, cornea or other refractive stromal opacity in the study eye affects retinal observation and examination.
3. Presence of ocular conditions that may affect suprachoroidal injection or the assessment of study endpoints.
4. Have undergone intraocular surgery in the study eye within 6 months.
5. Have received any gene therapy or cell therapy in the past.
6. Subjects with childbearing potential are unwilling to use contraceptive measures.
7. Presence of any of the following: active infection requiring systemic treatment which, in the opinion of the investigator, may affect the patient's participation or study results; positive hepatitis B surface antigen (HBsAg) with HBV DNA copy number > ULN; positive hepatitis C virus (HCV) antibody with HCV-RNA copy number > ULN; positive Treponema pallidum antibody; positive human immunodeficiency virus (HIV) antibody.
8. Diagnosis of malignancy within 5 years prior to screening (except for adequately treated carcinoma in situ of the cervix, basal cell or squamous cell skin cancer, or ductal carcinoma in situ of the breast after radical resection).
9. Suffering or having suffered from systemic immune system diseases.
10. Abnormal laboratory values considered clinically significant: alanine aminotransferase and/or aspartate aminotransferase >2.5×ULN, total bilirubin >1.5×ULN, serum creatinine >1.5×ULN, prothrombin time ≥1.5× ULN, activated partial thromboplastin time ≥1.5×ULN.
11. There is severe allergy or known allergy to the drugs used for treatment or examination in the research protocol, including allergy to study drugs.
12. Pregnant or lactating women; subjects of childbearing potential who are unable to use effective contraception from 2 weeks prior to screening until 6 months after administration.
13. Other circumstances that the researcher believes are not suitable for participating in this study

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety(Participants With Ocular and Non-ocular AEs (Adverse Events) and SAEs (Serious Adverse Events) | Baseline to day 7, day 14, month 1, 3, 6, 12
  The primary outcome measures are safety, determined by the number of ocular and non-ocular Study Drug-related adverse events (SDAE), treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs).

SECONDARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | Baseline to day 7, day 14, month 1, 2, 3, 6, 12
  Visual acuity of the study eye was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS)
Pigmentation of the Fundus | Baseline to day 7, day 14, month 1, 2, 3, 6, 12
  Evaluate retinal pigmentation and changes from baseline through fundus examination and fundus photography
Eye Movement | Baseline to month 1, 3, 6, 12
  The function of gaze, scanning, tracking and other movement
Macular Structure as Assessed by Swept Source Optical Coherence Tomography | Baseline to day 7, day 14, month 1, 2, 3, 6, 12
  Change in swept source optical coherence tomography(SS-OCT)
Electroretinogram | Baseline to month 1, 3, 6, 12
  The ERG measurement will be performed based on the standards of international society for clinical electrophysiology of vision (ISCEV)

OTHER OUTCOMES:
FST threshold | Baseline to month 1, 3, 6, 12
Contrast sensitivity, stereoscopic functional examination and color blindness examination | Baseline to month 1, 3, 6, 12
Structure and function of optic chiasm and visual pathway | Baseline to month 1, 3, 6 and 12
  Evaluate the structure and function of the optic chiasm and visual pathway of patients through visual evoked potential (VEP) and head MRI plain scan and functional imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Lu, Principal Investigator — Department of Ophthalmology, West China Hospital, Sichuan University
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China